CLINICAL TRIAL: NCT05796063
Title: Postoperative Gastric Point of Care Ultrasound (G-POCUS) in Abdominal Surgery: Can G-POCUS Guidance in Clinical Management of Gastrointestinal Recovery Lead to Better Outcomes?
Brief Title: Postoperative Gastric Point of Care Ultrasound (G-POCUS) in Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: iRISID-2022-1082
Record Dates: First submitted 2023-03-07; First posted 2023-04-03 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Ileus Postoperative; Postoperative Nausea and Vomiting
Keywords: gastric ultrasound; delayed bowel function; postoperative ileus
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): On postoperative day one, patients will be asked if they are having any GI symptoms. These are defined as presence of nausea, emesis, belching, and/or hiccups. In the intervention arm, clinicians will use the results of G-POCUS and presence/absence of GI symptoms to inform decision making according to one of two standardized algorithms.
  Interventions: Diagnostic Test: gastric point of care ultrasound
- Control (No Intervention): On postoperative day one, patients will be asked if they are having any GI symptoms. These are defined as presence of nausea, emesis, belching, and/or hiccups. In the control arm, presence of GI symptoms will be assessed, and once of two standardized algorithms which are representative of the current standard of care for postoperative diet management.

INTERVENTIONS:
Diagnostic Test: gastric point of care ultrasound — Patients will receive a gastric point of care ultrasound to evaluate for delayed gastric emptying. Gastric POCUS studies will be obtained using Kosmos, a handheld portable ultrasound that is FDA approved for clinical use. This product has already been validated for use, and this is not a novel application of the technology.
  Arms: Intervention

SUMMARY:
The purpose of this research is to determine if gastric point of care ultrasound (G-POCUS) can be used to help clinicians determine when to feed patients or when to insert or remove nasogastric tubes for patients recovering from colorectal or abdominal surgery.

Patients enrolled in the intervention group will have G-POCUS exams performed after surgery. The results of the exams will be used to make clinical decisions.

Researchers will compare these patients to patients receiving the usual care in the hospital after surgery.

DETAILED DESCRIPTION:
Delayed bowel function (DBF) and postoperative ileus (POI), or disruption of the normal forward peristaltic bowel activity after abdominal surgery are common complications in general surgery patients that can lead to nausea, emesis, bowel perforation, or aspiration pneumonitis. DBF and POI increase length of stay, morbidity, and mortality in general surgery patients. It is extremely difficult to predict who will develop DBF and POI. Further, diagnosing patients with postoperative DBF or POI is almost entirely based upon clinical acumen, history, and physical exam. To date no imaging or laboratory studies are specifically recommended to diagnose these complications.

Gastric Point of Care Ultrasound (G-POCUS) is a simple and reliable imaging modality that can be performed at the bedside and does not involve ionizing radiation. In the pilot study, it was hypothesized that G-POCUS volume (ie: whether a patient's stomach appears full or empty) would correlate with measures of delayed bowel functioning based on identification of full versus empty stomach postoperatively following colorectal surgery. We found that patients with full stomachs had a higher incidence of DBF, length of stay, emesis, and need for nasogastric tube (NGT) placement.

This will be a randomized single-blinded study of handheld G-POCUS in which the study population will be inpatients hospitalized after abdominal/colorectal surgery. Patients will be randomized to an unblinded intervention arm or an unblinded standard of care arm. On postoperative day 1 (POD1), patients will be asked if they are having any GI symptoms. These are defined as presence of nausea, emesis, belching, and/or hiccups. In the intervention arm, clinicians will use the results of G-POCUS and presence/absence of GI symptoms to inform decision making according to one of two standardized algorithms. In the control arm, presence of GI symptoms will be assessed, and once of two standardized algorithms which are representative of the current standard of care for postoperative diet management. Data from both groups will be used to determine if the G-POCUS studies' results can predict the incidence of primary or secondary outcomes (control) or if intervening on results of G-POCUS can decrease the incidence of undesirable outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Completed signed and dated informed consent form
  * Willing to comply with all study procedures
  * Male or female, 18 years of age or older
  * Presenting for a schedule elective colorectal/abdominal surgery, either open, robotic, or laparoscopic

Exclusion Criteria:

* History of gastroparesis or known gastric/intestinal motility disorder
* History of gastric/bariatric surgery
* Intubated/sedated postoperatively
* Presence of open abdominal wounds (including abdominal wound vac)
* Patients who received a complex abdominal wall reconstruction
* Class III/IV Wound (Contaminated/Infected/Dirty)
* Surgery was emergent/urgent/unscheduled
* NGT placed or present at time of operation
* Presence of ileostomy/colostomy
* J-pouch reconstruction patients
* Currently pregnant patients
* Patients aged <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Utility of G-POCUS as a clinical decision-making tool - diet advancement | post-operative day 1 until day of discharge from the hospital for patients in the intervention group
  Patients enrolled in the intervention arm will have G-POCUS exams performed. A previously validated algorithm will be used to determine if their stomach is full or empty. Based on this result, decisions by the clinical team will be made regarding the patients' diet, need for nasogastric decompression using a standardized algorithm.

SECONDARY OUTCOMES:
Utility of G-POCUS as a clinical decision-making tool - quality of care metrics | post-operative day 1 until day of discharge
  The results from the intervention group will be compared to the control group (which will also proceed according to a standardized algorithm that reflects the current standard of care) to determine if there are differences in length of stay and aspiration pneumonia/pneumonitis between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Phillips, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asgeirsson T, El-Badawi KI, Mahmood A, Barletta J, Luchtefeld M, Senagore AJ. Postoperative ileus: it costs more than you expect. J Am Coll Surg. 2010 Feb;210(2):228-31. doi: 10.1016/j.jamcollsurg.2009.09.028. Epub 2009 Nov 18. PMID 20113944
- [Background] Bragg D, El-Sharkawy AM, Psaltis E, Maxwell-Armstrong CA, Lobo DN. Postoperative ileus: Recent developments in pathophysiology and management. Clin Nutr. 2015 Jun;34(3):367-76. doi: 10.1016/j.clnu.2015.01.016. Epub 2015 Jan 31. PMID 25819420
- [Background] Gustafsson UO, Hausel J, Thorell A, Ljungqvist O, Soop M, Nygren J; Enhanced Recovery After Surgery Study Group. Adherence to the enhanced recovery after surgery protocol and outcomes after colorectal cancer surgery. Arch Surg. 2011 May;146(5):571-7. doi: 10.1001/archsurg.2010.309. Epub 2011 Jan 17. PMID 21242424
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Haskins SC, Kruisselbrink R, Boublik J, Wu CL, Perlas A. Gastric Ultrasound for the Regional Anesthesiologist and Pain Specialist. Reg Anesth Pain Med. 2018 Oct;43(7):689-698. doi: 10.1097/AAP.0000000000000846. PMID 30052550
- [Background] Heinberg EM, Finan MA, Chambers RB, Bazzett LB, Kline RC. Postoperative ileus on a gynecologic oncology service--do abdominal X-rays have a role? Gynecol Oncol. 2003 Jul;90(1):158-62. doi: 10.1016/s0090-8258(03)00247-6. PMID 12821357
- [Background] Lamm R, Collins M, Bloom J, Joel M, Iosif L, Park D, Reny J, Schultz S, Yeo CJ, Beausang D, Schwenk ES, Costanzo C, Phillips BR. Postoperative Handheld Gastric Point-of-Care Ultrasound and Delayed Bowel Function. J Am Coll Surg. 2023 Apr 1;236(4):554-559. doi: 10.1097/XCS.0000000000000536. Epub 2023 Jan 5. PMID 36602237
- [Background] Lamm R, Bloom J, Collins M, Goldman D, Beausang D, Costanzo C, Schwenk ES, Phillips B. A Role for Gastric Point of Care Ultrasound in Postoperative Delayed Gastrointestinal Functioning. J Surg Res. 2022 Aug;276:92-99. doi: 10.1016/j.jss.2022.02.028. Epub 2022 Mar 24. PMID 35339785
- [Background] Lamm R, Collins M, Bloom J, Joel M, Iosif L, Park D, Reny J, Schultz S, Phillips B, Schwenk E, Costanzo C. Novice User Learning Curve for Handheld Gastric Point of Care Ultrasound Evaluations to Detect Delayed Return of Postoperative Peristalsis. Am Surg. 2023 Dec;89(12):6290-6292. doi: 10.1177/00031348231156770. Epub 2023 Feb 14. No abstract available. PMID 36787243
- [Background] Mirbagheri N, Dunn G, Naganathan V, Suen M, Gladman MA. Normal Values and Clinical Use of Bedside Sonographic Assessment of Postoperative Gastric Emptying: A Prospective Cohort Study. Dis Colon Rectum. 2016 Aug;59(8):758-65. doi: 10.1097/DCR.0000000000000637. PMID 27384094
- [Background] Nielsen S, Degenhardt L, Hoban B, Gisev N. A synthesis of oral morphine equivalents (OME) for opioid utilisation studies. Pharmacoepidemiol Drug Saf. 2016 Jun;25(6):733-7. doi: 10.1002/pds.3945. Epub 2015 Dec 22. PMID 26693665
- [Background] Scarborough JE, Schumacher J, Kent KC, Heise CP, Greenberg CC. Associations of Specific Postoperative Complications With Outcomes After Elective Colon Resection: A Procedure-Targeted Approach Toward Surgical Quality Improvement. JAMA Surg. 2017 Feb 15;152(2):e164681. doi: 10.1001/jamasurg.2016.4681. Epub 2017 Feb 15. PMID 27926773
- [Background] Schwenk ES, Grant AE, Torjman MC, McNulty SE, Baratta JL, Viscusi ER. The Efficacy of Peripheral Opioid Antagonists in Opioid-Induced Constipation and Postoperative Ileus: A Systematic Review of the Literature. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):767-777. doi: 10.1097/AAP.0000000000000671. PMID 29016552
- [Background] Sommer NP, Schneider R, Wehner S, Kalff JC, Vilz TO. State-of-the-art colorectal disease: postoperative ileus. Int J Colorectal Dis. 2021 Sep;36(9):2017-2025. doi: 10.1007/s00384-021-03939-1. Epub 2021 May 11. PMID 33977334
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784
- [Background] Vather R, Trivedi S, Bissett I. Defining postoperative ileus: results of a systematic review and global survey. J Gastrointest Surg. 2013 May;17(5):962-72. doi: 10.1007/s11605-013-2148-y. Epub 2013 Feb 2. PMID 23377782
- [Background] Wu Z, Boersema GS, Dereci A, Menon AG, Jeekel J, Lange JF. Clinical endpoint, early detection, and differential diagnosis of postoperative ileus: a systematic review of the literature. Eur Surg Res. 2015;54(3-4):127-38. doi: 10.1159/000369529. Epub 2014 Dec 10. PMID 25503902
- [Background] Zhang X, Zheng W, Chen C, Kang X, Zheng Y, Bao F, Gan S, Zhu S. Goal-directed fluid therapy does not reduce postoperative ileus in gastrointestinal surgery: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Nov;97(45):e13097. doi: 10.1097/MD.0000000000013097. PMID 30407319